CLINICAL TRIAL: NCT06179160
Title: A Phase 1, Open-Label, Multicenter Study of INCB161734 in Participants With Advanced or Metastatic Solid Tumors With KRAS G12D Mutation
Brief Title: A Study to Evaluate INCB161734 in Participants With Advanced or Metastatic Solid Tumors With KRAS G12D Mutation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INCB161734-101; 2023-507091-47-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2023-12-12; First posted 2023-12-21 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumors
Keywords: INCB161734; KRASG12D Mutation; pancreatic ductal adenocarcinoma (PDAC); colorectal cancer (CRC); non-small cell lung cancer (NSCLC)
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab; Folfox protocol; IFL protocol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1a: Dose Escalation monotherapy (Experimental): INCB161734 at the protocol-defined dose strength based on cohort assignment.
  Interventions: Drug: INCB161734
- Part 1b: Dose Expansion monotherapy (Experimental): INCB161734 at the protocol-defined dose strength based on cohort assignment.
  Interventions: Drug: INCB161734
- Part 1c: Pharmacodynamic cohort (Experimental): INCB161734 at the protocol-defined dose strength based on cohort assignment.
  Interventions: Drug: INCB161734
- Part 2a: Dose Escalation combination (Experimental): INCB161734 in combination at the protocol-defined dose strength based on cohort assignment.
  Interventions: Drug: INCB161734; Drug: Cetuximab; Drug: Retifanlimab; Drug: GEMNabP; Drug: mFOLFIRINOX; Drug: FOLFOX; Drug: FOLFIRI; Drug: INCA33890
- Part 2b: Dose Expansion combination (Experimental): INCB161734 in combination at the protocol-defined dose strength based on cohort assignment.
  Interventions: Drug: INCB161734; Drug: Cetuximab; Drug: Retifanlimab; Drug: GEMNabP; Drug: mFOLFIRINOX; Drug: FOLFOX; Drug: FOLFIRI; Drug: INCA33890
- Part 1d: Food-Effect (Experimental): Evaluate food effect on drug exposure as defined in the protocol.
  Interventions: Drug: INCB161734

INTERVENTIONS:
Drug: INCB161734 — INCB161734 will be administered at protocol defined dose.
Drug: Cetuximab — Cetuximab will be administered at protocol defined dose.
  Arms: Part 2a: Dose Escalation combination; Part 2b: Dose Expansion combination
Drug: Retifanlimab — Retifanlimab will be administered at protocol defined dose.
  Arms: Part 2a: Dose Escalation combination; Part 2b: Dose Expansion combination
Drug: GEMNabP — GEMNabP will be administered at protocol defined dose.
  Arms: Part 2a: Dose Escalation combination; Part 2b: Dose Expansion combination
Drug: mFOLFIRINOX — mFOLFIRINOX will be administered at protocol defined dose.
  Arms: Part 2a: Dose Escalation combination; Part 2b: Dose Expansion combination
Drug: FOLFOX — FOLFOX will be administered at protocol defined dose.
  Arms: Part 2a: Dose Escalation combination; Part 2b: Dose Expansion combination
Drug: FOLFIRI — FOLFIRI will be administered at protocol defined dose.
  Arms: Part 2a: Dose Escalation combination; Part 2b: Dose Expansion combination
Drug: INCA33890 — INCA33890 will be administered at protocol defined dose.
  Arms: Part 2a: Dose Escalation combination; Part 2b: Dose Expansion combination

SUMMARY:
This study is conducted to determine the safety and tolerability of INCB161734 as a single agent or in combination with other anticancer therapies.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old.
* Locally advanced or metastatic solid tumor with KRAS G12D mutation.
* For Part 1a and Part 2 Combination Groups 1, 2, and 7: Disease progression on prior standard treatment, intolerance to or ineligibility for standard treatment, declined available therapies that are known to confer clinical benefit, or no standard available treatment to improve the disease outcome.
* Cohort specific requirements aas defined in the protocol.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

* Prior treatment with any KRAS G12D inhibitor
* Known additional invasive malignancy within 1 year of the first dose of study drug
* History of organ transplant, including allogeneic stem cell transplantation
* Significant, uncontrolled medical condition
* History or presence of an ECG abnormality
* Inadequate organ function

Other protocol-defined Inclusion/Exclusion Criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 710 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Dose Limiting Toxicities (DLTs) | Up to 28 days
  Dose-limiting toxicity will be defined as the occurrence of any of the toxicities as per protocol.
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to 2 years and 90 days
  Defined as adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug monotherapy and in combination with cetuximab and retifanlimab.
Number of participants with TEAEs leading to dose modification or discontinuation | Up to 2 years and 90 days
  Number of participants with TEAEs leading to dose modification or discontinuation.

SECONDARY OUTCOMES:
INCB161734 pharmacokinetic (PK) in Plasma | Up to approximately 90 days
  INCB161734 concentration in plasma.
Objective Response Rate (ORR) | Up to 2 years
  Defined as having a best overall Complete Response (CR) or Partial Response (PR), as determined by the investigator by radiographic disease assessment according to RECIST v1.1.
Disease Control Response (DCR) | Up to 2 years
  Defined as having a best overall response of CR, PR, or Stable Disease (SD) as determined by the investigator by radiographic disease assessment according to RECIST v1.1.
Duration of Response (DOR) | Up to 2 years
  Defined as the time from earliest date of disease response (Completed Response or Partial Response) until earliest date of disease progression as determined by the investigator by radiographic disease assessment according to RECIST v1.1 or death due to any cause if occurring sooner than progression.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (34):
- United States (13):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Stanford University, Palo Alto, California
  - UCLA Healthcare Hematology-Oncology, Santa Monica, California
  - Sarah Cannon Research Institue At Healthone, Denver, Colorado
  - Florida Cancer Specialists, Sarasota, Florida
  - Sidney Kimmel Comprehensive Cancer Center At Johns Hopkins, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Weill Cornell Medicine, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Jefferson University Hospitals, Philadelphia, Pennsylvania
  - Scri Oncology Partners, Nashville, Tennessee
  - Md Anderson Cancer Center, Houston, Texas
- Australia (5):
  - Chris Obrien Lifehouse, Camperdown, New South Wales
  - St Vincent'S Hospital Sydney, Darlinghurst, New South Wales
  - The Alfred Hospital, Melbourne, Victoria
  - Peter Maccallum Cancer Centre, North Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- Belgium (3):
  - Cliniques Universitaires Ucl Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen (Uza), Edegem
  - Universitair Ziekenhuis (Uz) Leuven, Leuven
- Canada (2):
  - The Ottawa Hospital Cancer Center, Ottawa, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
- France (3):
  - Centre Leon Berard, Lyon
  - Universitaire Du Cancer de Toulouse Institut Claudius Regaud Iuct-Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif
- Italy (3):
  - Fondazione Irccs Istituto Nazionale Dei Tumori, Milan
  - Irccs Istituto Clinico Humanitas, Rozzano
  - Centro Ricerche Cliniche Di Verona, Verona
- Japan (2):
  - National Cancer Center Hospital East, Chiba
  - The Cancer Institute Hospital of Jfcr, Tokyo
- Spain (3):
  - Hospital General Universitario Vall D Hebron, Barcelona
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Quironsalud Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study to Evaluate INCB161734 in Participants With Advanced or Metastatic Solid Tumors With KRAS G12D Mutation — https://incyteclinicaltrials.com/studies/incb161734-101